CLINICAL TRIAL: NCT03117699
Title: Continuation of the Exploration of the Standing Seated Passage of the Hemiplegic for the Realization of a New Transport Device
Brief Title: Seated - Standing Passage of the Hemiplegic
Acronym: PADH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 29BRC16.0012 PADH2
Record Dates: First submitted 2017-03-29; First posted 2017-04-18 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Hemiplegia
Keywords: Hemiplegia; transport device
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemiplegic subjects (Experimental): Testing of a new device for seated-standing passages after undergoing medical evaluation included Fugl Meyer scale, Berg scale and Bergego scale.
  Phase 1 :
  * 3 seated-standing passages with a handle equipped with 6 force captors
  * 3 seated-standing passages with the device
  Interventions: Device: New device for seated-standing passages
- Healthy volunteers (Experimental): Testing of a new device for seated-standing passages .
  Phase 1 :
  * 3 seated-standing passages without help
  * 3 seated-standing passages with a handle equipped with 6 force captors
  * 3 seated-standing passages with the device
  Interventions: Device: New device for seated-standing passages

INTERVENTIONS:
Device: New device for seated-standing passages — Phase 1 : The subject perform different seated-standing passages (see "Arm")
  Phase 2 : After being seated, the subject performs a course comprising:
  * A standing pass from sitting on a chair
  * A straight line movement
  * A succession of left and right turns
  * An upward and downward travel of less than 1%.
  * Standard doorway
  * Standing on the toilet
  * A sitting pass from the toilet
  * One way to a bed
  * A sitting pass on the bed
  * A passenger seat sitting upright from the bed
  * A return to the starting point
  * A sitting pass on the starting chair

SUMMARY:
This is a study for a new mechanical transport device adapted to the hemiplegic patients.

Healthy volunteers :

After explaining the protocol and presenting the movement laboratory, the subjects are equipped with reflective markers on the 4 limbs, the trunk and the head. The subjects are installed on a seat positioned in front of 2 force platforms installed on the ground. The seat is equipped with a force platform.

Phase 1 :

After being seated, the subject realizes :

* 3 seat to stand and stand to seat without assistance
* 3 seat to stand and stand to seat using a handle located in front of it (handle equipped with a 6-axis force sensor)
* 3 seat to stand and stand to seat using the experimental device This phase will last 45minutes (mn) (30mn of equipment and 15mn of sitting passengers standing)

Phase 2:

After being seated, the subject performs a course comprising:

* A standing pass from sitting on a chair
* A straight line movement
* A succession of left and right turns
* An upward and downward travel of less than 1%.
* Standard doorway
* Standing on the toilet
* A sitting pass from the toilet
* One way to a bed
* A sitting pass on the bed
* A passenger seat sitting upright from the bed
* A return to the starting point
* A sitting pass on the starting chair Each stage is timed. A subjective analysis of each step is done by a lickert scale on the perceived comfort and safety.

This phase 2 will last 30mn (15mn of course and 15mn of questions).

Hemiplegic subjects :

At each session, the subject is examined by a physician who evaluates the motor control (Fugl Meyer scale), the equilibrium (Berg scale) and the spatial hemineglect (Bergego scale).

Phase 1 is performed except the 3 seat to stand and stand to seat without assistance which are impossible.

Phase 2 is performed. An evaluation of the device over 4 hours is carried out for each subject in therapeutic apartment in simulated living conditions. The validation in living lab is carried out by an ergonomist and by a questionnaire on the comfort and safety of the various steps identified by the ergonomist.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers :

* aged 18-75 years
* Subject having given his consent
* Free from any neurological or cardiorespiratory locomotor pathology that may interfere with standing seated passages.

Hemiplegic patients :

* Left hemiplegia in one of the following groups :
* Walking with difficulty or not walking and able to stand with a stick or an armrest
* Walking difficult or not walking and unable to stand with a cane or an armrest.
* aged 18-90 years
* Subject having given his consent
* Subjects with a trunk balance to sit without support

Exclusion Criteria:

* aged less than 18 or more than 75 (healthy volunteers) or more than 90 (hemiplegic subjects)
* Pain during seated-standing passages
* Unstable medical condition
* Unable to consent
* Subject under legal protection
* Left-hemineglect making standing or seated (wheelchair) displacements impossible autonomously (for hemiplegic patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Time required to carry out each step of use of the device | Day 1
  Each step of phase 1 and phase 2 will be timed.

SECONDARY OUTCOMES:
Record of all adverse reactions. | Day 1
  The safety of the devices will be evaluated by the occurrence of adverse reactions.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Brest University Hospital, Brest
  - Centre de rééducation fonctionnelle de KERPAPE, Ploemeur

IPD SHARING:
Plan to Share IPD: No